CLINICAL TRIAL: NCT05808946
Title: The Effect of Alpha-Lipoic Acid on the Clinical Outcome of Patients With Sepsis
Brief Title: Alpha-Lipoic Acid in Patients With Sepsis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Lujayna AbdelAziz, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACUC-FP-ASURHDIRB2020110301158
Record Dates: First submitted 2023-03-19; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Sepsis
Keywords: Alpha Lipoic Acid; MCP-1; Mortality; Vasopressors; Efficacy; Safety
MeSH Terms: conditions — Sepsis | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha-Lipoic Acid Group (Experimental)
  Interventions: Drug: Alpha-Lipoic Acid; Drug: Sepsis Supportive Care
- Control Group (Active Comparator)
  Interventions: Drug: Sepsis Supportive Care

INTERVENTIONS:
Drug: Alpha-Lipoic Acid — 1200 mg of ALA daily (given as two 600 mg capsules once daily)
  Other Names: Thioctic Acid
  Arms: Alpha-Lipoic Acid Group
Drug: Sepsis Supportive Care — Appropriate IV fluid, Appropriate antibiotic, Vasopressors if needed, Mechanical ventilation if needed
  Other Names: Sepsis Management

SUMMARY:
Alpha-lipoic acid (ALA) is a powerful antioxidant that can help reduce the harmful effects of free radicals in the body. When the body is fighting sepsis, the immune response generates a lot of free radicals that can damage cells and tissues. ALA can neutralize these free radicals, reducing oxidative stress and preventing damage to cells and tissues.

ALA also has anti-inflammatory properties, meaning it can reduce inflammation in the body. Inflammation is a key feature of sepsis, and it can cause damage to organs and tissues. By reducing inflammation, ALA can help prevent damage to organs and tissues, reducing the risk of sepsis complications such as organ failure.

The objective of this research is to investigate the impact of ALA on individuals who have sepsis. The study will involve dividing the participants into two groups: a control group and an ALA group. The control group will receive the standard supportive care for sepsis management. Meanwhile, the ALA group will receive 1200 mg of ALA daily in addition to the standard care.

DETAILED DESCRIPTION:
Sepsis is considered a leading cause of death in hospitals and intensive care units (ICU) due to the body's excessive response to the invading pathogen, resulting in severe inflammation and oxidative stress. As a result, it is postulated that administering anti-inflammatory and antioxidant agents may have potential benefits on the clinical outcomes of patients with sepsis. Alpha-lipoic acid, a nutraceutical with both potent anti-inflammatory and antioxidant properties, could be a potential treatment option. Several animal models showed positive results when using ALA in septic rats. Hence, it might be a potential candidate for improving the clinical outcome in septic patients. Thus, the aim of this study is to evaluate the efficacy and safety of alpha-lipoic acid when administered at a dose of 1200 mg/day in septic patients.

This trial is a prospective randomized-controlled open label trial where a total number of 60 patients will be enrolled in the study. They will be randomized using simple randomization into the control group and the treatment group with a ratio of 1 to 1 (30 patients in each group). The control group will receive the standard supportive care of sepsis management. Supportive care typically involves a combination of interventions to stabilize the patient's condition and manage their symptoms such as administration of intravenous fluids (e.g.: normal saline) and appropriate antibiotics. Additionally, oxygen therapy, mechanical ventilation, and vasopressors (e.g.: norepinephrine or dobutamine) may be provided on an as-needed basis to support breathing and maintain blood pressure. Meanwhile, the ALA group will be given 1200 mg of ALA daily in addition to the standard care.

The efficacy of ALA will be assessed by tracking the mortality rates of enrolled patients during their hospital stay and 28 days after, as well as the duration of their ICU and hospital stay. The Sequential [Sepsis-related] Organ Failure Assessment (SOFA) score, C-reactive protein (CRP), Total Leukocytic Count (TLC), and plasma monocyte chemoattractant protein 1 (MCP-1) will also be measured at baseline and regularly during the study to evaluate ALA's impact on sepsis. Also, the need for mechanical ventilation and vasopressors will be recorded as an indicator of ALA's efficacy. The safety of ALA will be determined by monitoring the patients for any adverse effects that may occur due to the drug such as nausea or itching.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. Patients able to receive oral or enteral medication
3. Patients with confirmed diagnosis of sepsis according to Sepsis-3 definition; documented or suspected infection associated with organ dysfunction identified by acute change in total SOFA score of 2 points or more.

Exclusion Criteria:

1. Patients with septic shock defined as patients with sepsis who has persistent hypotension that necessitates the use of vasopressors to maintain MAP greater than or equal to 65mmHg and a blood lactate level greater than 2 mmol/L (18 mg/dL) despite absence of hypovolemia.
2. Patients on mechanical ventilation at baseline.
3. Pregnant women
4. Patients already receiving ALA supplementation before ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days since patient enrollment in the study
  The patient will be followed-up for mortality rate during hospital stay and up to 28 days.

SECONDARY OUTCOMES:
Plasma MCP-1 | Plasma samples will be collected on days 1, 3 and 7 for each patient enrolled
  Monocyte chemoattractant protein-1 (MCP-1) will be assessed in each patient as an inflammatory marker.
SOFA score | Assessed on day 1, 3 and 7 and then every 3 days till patient is discharged or death occurs, up to maximum 28 days.
  A scoring system used to measure the extent of organ dysfunction/failure in critically ill patients. The score is calculated based on six different parameters: respiratory (PaO2/FiO2 ratio), cardiovascular (mean arterial pressure (MAP)), hepatic (serum bilirubin level), coagulation (platelet count), renal (serum creatinine level and urine output), and neurological (Glasgow Coma Scale).
  This makes the SOFA score a composite outcome.
Length of ICU stay | 28 days
  The total duration of ICU stay will be estimated for each patient.
Length of hospital stay | 28 days
  The total duration of hospital stay will be estimated for each patient.
Need for Mechanical Ventilation | 28 days
  Number of patients requiring mechanical ventilation will be recorded along with the duration of ventilation
Need for Vasopressors | 28 days
  Number of patients requiring vasopressors as norepinephrine or dopamine will be recorded along with the dose and the duration of vasopressor administration
Adverse Effects of Alpha-Lipoic Acid | 28 days
  All adverse effects experienced by the participants will be recorded in both arms. Expected side effects include gastrointestinal side effects (e.g.: nausea and vomiting) and hypersensitivity of the skin (e.g.: urticaria and itching sensation).

CONTACTS AND LOCATIONS:
Overall Officials: Lujayna M AbdelAziz, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Specialized Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soltani R, Alikiaie B, Shafiee F, Amiri H, Mousavi S. Coenzyme Q10 improves the survival and reduces inflammatory markers in septic patients. Bratisl Lek Listy. 2020;121(2):154-158. doi: 10.4149/BLL_2020_022. PMID 32115970
- [Background] Zhu T, Liao X, Feng T, Wu Q, Zhang J, Cao X, Li H. Plasma Monocyte Chemoattractant Protein 1 as a Predictive Marker for Sepsis Prognosis: A Prospective Cohort Study. Tohoku J Exp Med. 2017 Feb;241(2):139-147. doi: 10.1620/tjem.241.139. PMID 28202856
- [Background] Lowes DA, Webster NR, Murphy MP, Galley HF. Antioxidants that protect mitochondria reduce interleukin-6 and oxidative stress, improve mitochondrial function, and reduce biochemical markers of organ dysfunction in a rat model of acute sepsis. Br J Anaesth. 2013 Mar;110(3):472-80. doi: 10.1093/bja/aes577. Epub 2013 Feb 4. PMID 23381720
- [Background] Salehi B, Berkay Yilmaz Y, Antika G, Boyunegmez Tumer T, Fawzi Mahomoodally M, Lobine D, Akram M, Riaz M, Capanoglu E, Sharopov F, Martins N, Cho WC, Sharifi-Rad J. Insights on the Use of alpha-Lipoic Acid for Therapeutic Purposes. Biomolecules. 2019 Aug 9;9(8):356. doi: 10.3390/biom9080356. PMID 31405030
- [Background] Park S, Karunakaran U, Jeoung NH, Jeon JH, Lee IK. Physiological effect and therapeutic application of alpha lipoic acid. Curr Med Chem. 2014;21(32):3636-45. doi: 10.2174/0929867321666140706141806. PMID 25005184
- [Background] Dewi Perwito Sari, I.S.a.J.K., THE MECHANISM OF ALA ON REDUCING THE MDA LEVEL AND MCP-1 EXPRESSION IN ENDOTHELIAL DYSFUNCTION OF HYPERCHOLESTEROLEMIA RAT MODEL. Folia Medica Indonesiana, 2016. 52.
- [Background] Rius-Perez S, Torres-Cuevas I, Millan I, Ortega AL, Perez S. PGC-1alpha, Inflammation, and Oxidative Stress: An Integrative View in Metabolism. Oxid Med Cell Longev. 2020 Mar 9;2020:1452696. doi: 10.1155/2020/1452696. eCollection 2020. PMID 32215168
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Tibullo D, Li Volti G, Giallongo C, Grasso S, Tomassoni D, Anfuso CD, Lupo G, Amenta F, Avola R, Bramanti V. Biochemical and clinical relevance of alpha lipoic acid: antioxidant and anti-inflammatory activity, molecular pathways and therapeutic potential. Inflamm Res. 2017 Nov;66(11):947-959. doi: 10.1007/s00011-017-1079-6. Epub 2017 Jul 4. PMID 28676917
- [Result] Mendoza-Nunez VM, Garcia-Martinez BI, Rosado-Perez J, Santiago-Osorio E, Pedraza-Chaverri J, Hernandez-Abad VJ. The Effect of 600 mg Alpha-lipoic Acid Supplementation on Oxidative Stress, Inflammation, and RAGE in Older Adults with Type 2 Diabetes Mellitus. Oxid Med Cell Longev. 2019 Jun 12;2019:3276958. doi: 10.1155/2019/3276958. eCollection 2019. PMID 31285784
- [Result] Gomes MB, Negrato CA. Alpha-lipoic acid as a pleiotropic compound with potential therapeutic use in diabetes and other chronic diseases. Diabetol Metab Syndr. 2014 Jul 28;6(1):80. doi: 10.1186/1758-5996-6-80. eCollection 2014. PMID 25104975
- [Result] Dworacka M, Iskakova S, Krzyzagorska E, Wesolowska A, Kurmambayev Y, Dworacki G. Alpha-lipoic acid modifies circulating angiogenic factors in patients with type 2 diabetes mellitus. Diabetes Res Clin Pract. 2015 Feb;107(2):273-9. doi: 10.1016/j.diabres.2014.11.005. Epub 2014 Dec 3. PMID 25511715
- [Result] Jia J, Gong X, Zhao Y, Yang Z, Ji K, Luan T, Zang B, Li G. Autophagy Enhancing Contributes to the Organ Protective Effect of Alpha-Lipoic Acid in Septic Rats. Front Immunol. 2019 Jul 2;10:1491. doi: 10.3389/fimmu.2019.01491. eCollection 2019. PMID 31333648
- [Result] Petronilho F, Florentino D, Danielski LG, Vieira LC, Martins MM, Vieira A, Bonfante S, Goldim MP, Vuolo F. Alpha-Lipoic Acid Attenuates Oxidative Damage in Organs After Sepsis. Inflammation. 2016 Feb;39(1):357-365. doi: 10.1007/s10753-015-0256-4. PMID 26431839
- [Result] Hiller S, DeKroon R, Xu L, Robinette J, Winnik W, Alzate O, Simington S, Maeda N, Yi X. alpha-Lipoic acid protects mitochondrial enzymes and attenuates lipopolysaccharide-induced hypothermia in mice. Free Radic Biol Med. 2014 Jun;71:362-367. doi: 10.1016/j.freeradbiomed.2014.03.022. Epub 2014 Mar 24. PMID 24675228
- [Result] Della Giustina A, Goldim MP, Danielski LG, Florentino D, Mathias K, Garbossa L, Oliveira Junior AN, Fileti ME, Zarbato GF, da Rosa N, Martins Laurentino AO, Fortunato JJ, Mina F, Bellettini-Santos T, Budni J, Barichello T, Dal-Pizzol F, Petronilho F. Alpha-lipoic acid attenuates acute neuroinflammation and long-term cognitive impairment after polymicrobial sepsis. Neurochem Int. 2017 Sep;108:436-447. doi: 10.1016/j.neuint.2017.06.003. Epub 2017 Jun 10. PMID 28606823
- [Result] Jiang S, Zhu W, Li C, Zhang X, Lu T, Ding Z, Cao K, Liu L. alpha-Lipoic acid attenuates LPS-induced cardiac dysfunction through a PI3K/Akt-dependent mechanism. Int Immunopharmacol. 2013 May;16(1):100-7. doi: 10.1016/j.intimp.2013.03.024. Epub 2013 Apr 3. PMID 23562296
- [Result] Koh EH, Lee WJ, Lee SA, Kim EH, Cho EH, Jeong E, Kim DW, Kim MS, Park JY, Park KG, Lee HJ, Lee IK, Lim S, Jang HC, Lee KH, Lee KU. Effects of alpha-lipoic Acid on body weight in obese subjects. Am J Med. 2011 Jan;124(1):85.e1-8. doi: 10.1016/j.amjmed.2010.08.005. PMID 21187189
- [Result] Kim BJ, Hunter A, Brucker AJ, Hahn P, Gehrs K, Patel A, Edwards AO, Li Y, Khurana RN, Nissim I, Daniel E, Grunwald J, Ying GS, Pistilli M, Maguire MG, Dunaief JL. Orally Administered Alpha Lipoic Acid as a Treatment for Geographic Atrophy: A Randomized Clinical Trial. Ophthalmol Retina. 2020 Sep;4(9):889-898. doi: 10.1016/j.oret.2020.03.019. Epub 2020 Apr 2. PMID 32418846